CLINICAL TRIAL: NCT03016520
Title: An Open-label, Randomized, Single-dose, 2-way Crossover Study to Compare the Pharmacokinetics and Safety of DWJ1392 and DWC20164 in Healthy Male Volunteers
Brief Title: Pharmacokinetics and Safety Study of DWJ1392 and DWC20164 in Healthy Male Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DW_DWJ1392001
Record Dates: First submitted 2017-01-09; First posted 2017-01-10 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-01

CONDITIONS: Healthy

ARMS (2):
- Test drug (Experimental): DWJ1392
  Interventions: Drug: DWJ1392
- Reference drug (Experimental): DWC20164
  Interventions: Drug: DWC20164

INTERVENTIONS:
Drug: DWJ1392
  Arms: Test drug
Drug: DWC20164
  Arms: Reference drug

SUMMARY:
The purpose of this study to Compare the safety and pharmacokinetics of DWJ1392 and DWC20164 in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant findings
* Age 19-50 years at screening

Exclusion Criteria:

* Who has allergy to investigational product

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2017-01-09 (Actual); Primary Completion 2017-01-26 (Actual); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | 0-72 hours
Area under the plasma concentration versus time curve (AUC) | 0-72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul ST. Mary's Hospital, Seoul, South Korea